CLINICAL TRIAL: NCT04742452
Title: Comparison of Partial Rotator Cuff Repair vs. Superior Capsular Reconstruction for Irreparable Rotator Cuff Tears
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Lake Health (Unknown); Midwest Orthopaedics at Rush (Other)
Responsible Party: Principal Investigator, Robert J. Gillespie, Chief, Shoulder and Elbow Surgery, UH Cleveland Medical Center Program Director, Orthopaedic Surgery, UH Cleveland Medical Center Associate Professor, CWRU School of Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20201107
Record Dates: First submitted 2020-12-10; First posted 2021-02-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Rotator Cuff Tears
Keywords: Superior capsular reconstruction; Partial rotator cuff repair; Magnetic resonance imaging
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superior Capsular Reconstruction (Active Comparator)
  Interventions: Procedure: Superior Capusular Reconstruction
- Partial Rotator Cuff Repair (Placebo Comparator)
  Interventions: Procedure: Partial Rotator Cuff Repair

INTERVENTIONS:
Procedure: Superior Capusular Reconstruction — Superior capsular reconstruction is one treatment option for massive and irreparable rotator cuff tears. The superior shoulder capsule, a thin membranous structure located on the inferior surface of the supraspinatus and infraspinatus muscles, is often torn in this type of rotator cuff tear. In superior capsular reconstruction, this structure is reconstructed with acellular dermal allograft.
  Arms: Superior Capsular Reconstruction
Procedure: Partial Rotator Cuff Repair — Partial rotator cuff repair can be performed, in conjunction with other procedures such as subacromial decompression and biceps tenodesis, when a rotator cuff tear is not amenable to a complete repair.
  Arms: Partial Rotator Cuff Repair

SUMMARY:
The primary objective of this prospective randomized controlled trial is to compare pain and functional outcomes between two surgical modalities for irreparable rotator cuff tears as measured by the pain visual analog scale (VAS), simple shoulder test (SST), American Shoulder and Elbow Surgery shoulder score (ASES), and Patient Reported Outcomes Measurement Information System (PROMIS) 29 score at 6 weeks, 3, 6, 12, and 24 months post-operatively. The two surgical modalities of interest are partial rotator cuff repair alone and partial rotator cuff repair with superior capsule reconstruction (SCR). The secondary objective of this study is determine the failure rate of partial repair alone vs. partial repair with SCR via magnetic resonance imaging (MRI) at 12 months post-operatively. The information gained from this investigation will be useful to discern if SCR provides any benefit to patients with irreparable rotator cuff tears. The investigators hypothesize that there is no statistically significant difference in pain and functional outcomes between partial rotator cuff repair alone versus partial rotator cuff repair with SCR. In addition, the investigators hypothesize that the failure rate will be significantly higher in patients undergoing partial rotator cuff repair with SCR.

DETAILED DESCRIPTION:
Rotator cuff injury is a commonly encountered problem within the United States. In most cases, surgical repair can reduce pain and restore baseline functional status. However, in the case of an irreparable rotator cuff tear, management becomes more challenging as these injuries tend to be larger in size, are inelastic secondary to tendon retraction, and exhibit fatty infiltration and rotator cuff atrophy1. A multitude of surgical approaches for an irreparable rotator cuff tear have been described in the literature, including partial repair alone, partial repair with superior capsular reconstruction (SCR), arthroscopic debridement, graft interposition, balloon spacer arthroplasty, tendon transfers, and reverse total shoulder arthroplasty (rTSA)2. In younger patients, the traditional approach to managing these injuries involved partial rotator cuff repair with subacromial decompression and debridement with the hopes of providing the patient with some restoration of function and pain relief3,4. Clinical studies have demonstrated that partial repair can lead to an improvement in pain and function in the early post-operative period; long-term outcomes following this procedure were less reliable3. In addition, a high rate of failure has been associated with partial rotator cuff repair alone. Partial repair with SCR is a relatively new surgical procedure that has become an increasingly popular treatment modality in recent years because of early promising biomechanical and functional outcomes5,6. However, there have been no prospective randomized assessments of SCR. Therefore, the long-term outcomes of SCR compared to the standard of care, namely partial rotator cuff repair, are unknown.

This will be a multi-center, prospective randomized controlled trial. Prior to enrollment, patients will be screened for inclusion criteria. Participants who meet the eligibility criteria and are suspected to have an irreparable rotator cuff tear will be randomized into one of the two treatment arms prior to surgery. Group 1 will receive partial rotator cuff repair alone while group 2 will receive partial rotator cuff repair with SCR. All patients with suspected irreparable rotator cuff tears will be consented in clinic. There is the potential situation where the surgeon believed that the rotator cuff tear was irreparable based on clinical and radiographic evidence but was able to completely repair the tear intraoperatively. Based on the modified intention-to-treat (mITT) principle, these select patients will be dropped from the study and will no longer be followed for research purposes. Randomization will occur with a stratified randomization excel spreadsheet. Each group will be followed post-operatively for 24 months. The primary objective of this study is to compare pain and functional outcomes between the two treatment arms. The secondary objective is to assess the failure rate between the two treatment arms.

Study Procedures

1. All patients with a strongly suspected irreparable rotator cuff tear will be identified in the clinics of the treating physicians and be screened for inclusion and exclusion criteria. The consent form will be reviewed in depth with the patients by an IRB-approved member of the study team, and all questions will be answered prior to enrollment in the study. Patients will be asked if they need additional time to review the consent, and no coercion will occur throughout the consent process. Although patients will be consented at this clinic visit, they will be informed that there is a possibility that they will ultimately be excluded from the study because an irreparable rotator cuff tear can only be confirmed intraoperatively.
2. At the initial pre-operative clinic visit, patient demographics will be collected and the pain and functional status of patients will be assessed using VAS, SST, ASES, and PROMIS-29 scores. It should take approximately 15 minutes to complete these surveys in clinic.
3. Patients requiring medical clearance to ensure their health is optimized for surgery will do so. After receiving medical clearance (if needed), the patients will undergo surgery.
4. Patients will be randomized prior to surgery into one of two possible treatment arms as described above. Stratified randomization will be performed with Microsoft Excel. If a patient, who was suspected to have an irreparable rotator cuff tear based on clinical and radiographic findings, is amenable to a complete rotator cuff tear, they will be dropped from the study and no longer followed for research purposes. This is based on the mITT principle.
5. On the day of surgery, the patient will receive either a partial rotator cuff repair alone or a partial rotator cuff repair with SCR.
6. Intraoperative data will be collected. For both groups, the investigators will assess if the following were performed during the procedure: subacromial decompression, biceps tenotomy vs. tenodesis, marginal convergence, single vs. double-row repair, and repair of the subscapularis muscle. For the SCR group, the size (mm2) and width (mm) of the acellular dermal allograft will be recorded. Finally, any complications that occur intraoperatively will be recorded for both groups.
7. After discharge from the surgery center, both groups of patients will be given identical pain medication regimens, post-operative restrictions, and clinical follow-up schedule. They will be instructed to follow-up in clinic at 6 weeks, 3, 6, 12, and 24 months post-operatively.
8. At each post-operative appointment, the patients will again be administered the VAS, SST, ASES, and PROMIS-29 questionnaires. Complications will be assessed at each visit. In addition, at the 12-month follow-up appointment, each patient in both groups will be given a prescription for an MRI of the operative shoulder to assess for failure of the repair.
9. Key variables for analysis will be found within the electronic medical record, and in questionnaires administered at clinic appointments. They include: age at time of surgery, sex, height, weight, hand dominance, laterality of surgery, mechanism of injury, and surgical complications (e.g., infection, failure of repair).

ELIGIBILITY:
Inclusion Criteria:

* Age range: ≥18 years
* Irreparable rotator cuff tear suspected on pre-operative MRI

Exclusion Criteria:

* Pregnant, illiterate, or non-English speaking individuals
* Rotator cuff pathology amenable to a complete repair intraoperatively
* Moderate to severe rotator cuff arthropathy (Hamada grade ≥3)
* Presence of glenohumeral arthritis on radiographs
* Irreparable subscapularis muscle intraoperatively
* Active infection within the ipsilateral glenohumeral joint
* Neurologic pathology limiting shoulder function
* Current smoker
* Workers' compensation claim

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analog Scale (VAS) | 6 weeks
  Scale of 0 to 10; 0 is no pain, 10 is the most amount of pain
Pain Visual Analog Scale (VAS) | 3 months
  Scale of 0 to 10; 0 is no pain, 10 is the most amount of pain
Pain Visual Analog Scale (VAS) | 6 months
  Scale of 0 to 10; 0 is no pain, 10 is the most amount of pain
Pain Visual Analog Scale (VAS) | 12 months
  Scale of 0 to 10; 0 is no pain, 10 is the most amount of pain
Pain Visual Analog Scale (VAS) | 24 months
  Scale of 0 to 10; 0 is no pain, 10 is the most amount of pain
American Shoulder and Elbow Society (ASES) score | 6 weeks
  Minimum score is 0, Maximum score is 100; 50% weighted for pain, 50% weighted for function. The higher the number the better the outcome.
American Shoulder and Elbow Society (ASES) score | 3 months
  Minimum score is 0, Maximum score is 100; 50% weighted for pain, 50% weighted for function. The higher the number the better the outcome.
American Shoulder and Elbow Society (ASES) score | 6 months
  Minimum score is 0, Maximum score is 100; 50% weighted for pain, 50% weighted for function. The higher the number the better the outcome.
American Shoulder and Elbow Society (ASES) score | 12 months
  Minimum score is 0, Maximum score is 100; 50% weighted for pain, 50% weighted for function. The higher the number the better the outcome.
American Shoulder and Elbow Society (ASES) score | 24 months
  Minimum score is 0, Maximum score is 100; 50% weighted for pain, 50% weighted for function. The higher the number the better the outcome.
Simple Shoulder Test (SST) | 6 weeks
  Minimum score is 0%, maximum is 100%. 12 yes/no questions. Higher scores correspond with better outcomes.
Simple Shoulder Test (SST) | 3 months
  Minimum score is 0%, maximum is 100%. 12 yes/no questions. Higher scores correspond with better outcomes.
Simple Shoulder Test (SST) | 6 months
  Minimum score is 0%, maximum is 100%. 12 yes/no questions. Higher scores correspond with better outcomes.
Simple Shoulder Test (SST) | 12 months
  Minimum score is 0%, maximum is 100%. 12 yes/no questions. Higher scores correspond with better outcomes.
Simple Shoulder Test (SST) | 24 months
  Minimum score is 0%, maximum is 100%. 12 yes/no questions. Higher scores correspond with better outcomes.
Patient Reported Outcomes Measurement Information Systems (PROMIS)-29 | 6 weeks
  29 question form. Scores range from 0 to 100. Higher scores correspond with better outcomes. Questions assess physical function, anxiety, depression, fatigue, pain interference, sleep quality, and social activity.
Patient Reported Outcomes Measurement Information Systems (PROMIS)-29 | 3 months
  29 question form. Scores range from 0 to 100. Higher scores correspond with better outcomes. Questions assess physical function, anxiety, depression, fatigue, pain interference, sleep quality, and social activity.
Patient Reported Outcomes Measurement Information Systems (PROMIS)-29 | 6 months
  29 question form. Scores range from 0 to 100. Higher scores correspond with better outcomes. Questions assess physical function, anxiety, depression, fatigue, pain interference, sleep quality, and social activity.
Patient Reported Outcomes Measurement Information Systems (PROMIS)-29 | 12 months
  29 question form. Scores range from 0 to 100. Higher scores correspond with better outcomes. Questions assess physical function, anxiety, depression, fatigue, pain interference, sleep quality, and social activity.
Patient Reported Outcomes Measurement Information Systems (PROMIS)-29 | 24 months
  29 question form. Scores range from 0 to 100. Higher scores correspond with better outcomes. Questions assess physical function, anxiety, depression, fatigue, pain interference, sleep quality, and social activity.

SECONDARY OUTCOMES:
Graft/repair integrity via magnetic resonance imaging | 12-months post-operatively.
  Assessing the integrity of the repair, either SCR or the partial repair, to see if it is still intact at 12 months post-operatively.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Lake Health, Willoughby, Ohio

REFERENCES:
- [Background] Bedi A, Dines J, Warren RF, Dines DM. Massive tears of the rotator cuff. J Bone Joint Surg Am. 2010 Aug 4;92(9):1894-908. doi: 10.2106/JBJS.I.01531. PMID 20686065
- [Background] Carver TJ, Kraeutler MJ, Smith JR, Bravman JT, McCarty EC. Nonarthroplasty Surgical Treatment Options for Massive, Irreparable Rotator Cuff Tears. Orthop J Sports Med. 2018 Nov 7;6(11):2325967118805385. doi: 10.1177/2325967118805385. eCollection 2018 Nov. PMID 30480007
- [Background] Cvetanovich GL, Waterman BR, Verma NN, Romeo AA. Management of the Irreparable Rotator Cuff Tear. J Am Acad Orthop Surg. 2019 Dec 15;27(24):909-917. doi: 10.5435/JAAOS-D-18-00199. PMID 31206436
- [Background] Walch G, Edwards TB, Boulahia A, Nove-Josserand L, Neyton L, Szabo I. Arthroscopic tenotomy of the long head of the biceps in the treatment of rotator cuff tears: clinical and radiographic results of 307 cases. J Shoulder Elbow Surg. 2005 May-Jun;14(3):238-46. doi: 10.1016/j.jse.2004.07.008. PMID 15889020
- [Background] Denard PJ, Brady PC, Adams CR, Tokish JM, Burkhart SS. Preliminary Results of Arthroscopic Superior Capsule Reconstruction with Dermal Allograft. Arthroscopy. 2018 Jan;34(1):93-99. doi: 10.1016/j.arthro.2017.08.265. Epub 2017 Nov 13. PMID 29146165
- [Background] Mihata T, Lee TQ, Watanabe C, Fukunishi K, Ohue M, Tsujimura T, Kinoshita M. Clinical results of arthroscopic superior capsule reconstruction for irreparable rotator cuff tears. Arthroscopy. 2013 Mar;29(3):459-70. doi: 10.1016/j.arthro.2012.10.022. Epub 2013 Jan 28. PMID 23369443